CLINICAL TRIAL: NCT00971854
Title: Alteration of Deep Brain Stimulation Parameters for Dystonia- A Double Blinded Randomised Controlled Trial
Brief Title: Alteration of Deep Brain Stimulation Parameters for Dystonia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Heather House, University of Oxford
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09/H0603/11; R&D Study - 5898
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-09

CONDITIONS: Dystonia
Keywords: Dystonia
MeSH Terms: conditions — Dystonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 60 Hz stimulation (Experimental): Experimental reduced frequency pallidal stimulation
  Interventions: Procedure: Alteration of deep brain stimulator settings
- 130 Hz stimulation (No Intervention): Current standard pallidal stimulation setting
  Interventions: Procedure: Alteration of deep brain stimulator settings

INTERVENTIONS:
Procedure: Alteration of deep brain stimulator settings — From 130Hz to 60Hz pallidal stimulation

SUMMARY:
Deep brain stimulation (DBS) involves placing electrodes into the brain. Through these electrodes, artificial electrical signals are chronically delivered into deep brain regions in order to alter abnormal brain activity. The artificial electrical signals are generated by a battery that is inserted under the skin of the chest. DBS is used to treat several disorders of movement, including dystonia. In dystonia, the electrodes are inserted into a brain region called the globus pallidus.

Globus pallidus stimulation can be very effective therapy for dystonia. However not all patients are equally responsive and therapeutic outcomes can be frustratingly variable. The reason for this variability is unclear. Such variability in response may need to be met by tailoring stimulation to individual patients.

Another issue with deep brain stimulation is battery life. Eventually, batteries become depleted and need to be replaced. Such battery replacements require an operation, hospital stay and the risk of introducing infection. The high electrical energy that has been used to treat dystonia means that batteries are typically replaced every year or two.

The artificial electrical signals of deep brain stimulation are delivered with three parameters; frequency (Hertz - Hz), voltage (volts) and pulse width (microseconds). It has recently been reported that lower frequency stimulation, at 60Hz rather than 130Hz, can be used effectively to treat dystonia. Such 60Hz stimulation may be more effective for some patients than others. The lower energy demands of 60Hz stimulation would also greatly improve battery life (potentially doubling battery life).

The aim of this study is to assess if 60Hz stimulation is more effective in ameliorating the dystonia of patients who have responded poorly to 130Hz pallidal stimulation. The current status of the evidence is one of clinical equipoise (uncertainty) and therefore suits a double blinded randomised trial.

ELIGIBILITY:
Inclusion Criteria:

* Primary dystonia (focal cervical or generalised dystonia) who are receiving chronic (>1 year) bilateral pallidal stimulation but have had poor therapeutic responses (< 50% improvement in relevant dystonia severity rating scale*) despite confirmation of accurate electrode position.
* Able to understand study requirements - able to provide consent.

  * Relevant dystonia rating scales: Cervical dystonia - severity subsection of the Toronto Western Hospital spasmodic torticollis rating scale; Generalised dystonia - severity section of the Burke Fahn Marsden rating scale.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-01 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
To assess if the stimulation frequency of 60 Hz is superior to 130 Hz for patients with primary dystonia who have responded poorly to standard 130 Hz pallidal stimulation | 6 months

SECONDARY OUTCOMES:
Assess any potential changes in anxiety, mood, cognition | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tipu Aziz, Professor, Principal Investigator — University of Oxford, Nuffield Department of Surgery
Locations (1):
- University of Oxford, Nuffield Department of Surgery, Oxford, Oxfordshire, United Kingdom